CLINICAL TRIAL: NCT00841386
Title: Treatment of Keratoconus Using Collagen Cross-Linking By Means of Topical Riboflavin and UV Light.
Brief Title: Treatment of Keratoconus Using Collagen Cross-Linking
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University at Buffalo (Other)
Responsible Party: James J. Reidy, M.D., Department of Ophthalmology, SUNY at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101365
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-01

CONDITIONS: Keratoconus
Keywords: Cornea; Keratoconus; Ectasia; Riboflavin; Collagen cross-linking
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Dilatation, Pathologic | interventions — Flavin Mononucleotide; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cross-linking treatment (Experimental): Topical anesthesia (lidocaine jelly 2%) will be used. The central 9 mm of corneal epithelium will be removed cautiously with an Amoils brush. Riboflavin 0.1% solution will be applied (10 mg riboflavin-5-phosphate in 10 ml dextran T-500 20% solution, supplied in a sterile, single dose container) to the cornea every 2-3 minutes for 15 minutes and then every 5 minutes thereafter. The UV source will be from the CBM VEGA X-linker (CSO, Florence, Italy). A wavelength of 370 nm will be used to direct 5.4 J/cm2 to the area of cornea debrided for 30 minutes. The distance from the UV source to the cornea will be 1.5 to 5.4 cm.
  Interventions: Drug: Riboflavin-5-phosphate
- Sham treatment group (Sham Comparator): Topical anesthesia (lidocaine jelly 2%) will be used. Differing from the treatment group, no epithelium will be debrided, but instead, this step will be skipped and a 2% methylcellulose solution combined with 1% fluorescein dye will be applied to the cornea every 5 minutes for 30 minutes. The patient will be placed under the UV device, but instead of the UV light, the LED aiming beam will be applied for 30 minutes.
  Interventions: Drug: Sham cross-linking

INTERVENTIONS:
Drug: Riboflavin-5-phosphate — Riboflavin 0.1% (10 mg riboflavin-5-phosphate in 10 ml dextran T-500 20% solution, supplied in a sterile, single dose container) will be applied to the cornea every 2-3 minutes for 15 minutes prior to starting UV irradiation. The UV irradiation will be given in six 5 minute intervals. Additional riboflavin will be administered following each 5 minute UV treatment.
  Other Names: Ricrolin (SOOFT Italia Inc.)
  Arms: Cross-linking treatment
Drug: Sham cross-linking — Topical anesthesia (lidocaine jelly 2%) will be used. Differing from the treatment group, no epithelium will be debrided, but instead, this step will be skipped and 2% methylcellulose solution with 1% sodium fluorescein will be applied to the cornea every 5 minutes for 15 minutes, and then every 5 minutes during the sham UV treatment. The patient will be placed under the UV device, and the aiming beam applied.
  Other Names: Goniosol
  Arms: Sham treatment group

SUMMARY:
The purpose of this study is to determine the effectiveness of collagen cross-linking in the cornea in halting the progression and possibly partially reversing the effects of keratoconus. Keratoconus is a progressive weakening in the cornea that causes irregular astigmatism and thinning of the cornea. The overall effect is reduction of vision, and in more advanced cases, scarring of the cornea that may lead to the need for corneal transplantation. Cross-linking has been shown increase the rigidity of the cornea. The patients would be treated once and then followed over 24 months. .

DETAILED DESCRIPTION:
The goal is for two groups of approximately 66 patients to be included in the study. One eye from the first group will undergo treatment, while the second group of age matched individuals will serve as a control. It will be a prospective, randomized, blinded study. Each patient will be randomized at the beginning of enrollment in the study and will receive a randomization number. The following parameters will be followed: 1. Best corrected spectacle acuity (BCSA) 2. The steepest keratometry measurement (KMax) as measured by computerized corneal topography 3. Apical corneal thickness 4. Corneal mechanical resistance. These measurements will be repeated at 1 month, 3 months, 6 months, 12, 18, and 24 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* no prior history of ocular surgery
* treatment eye must have a maximum corneal power of between 47 D and 60 diopters
* corneal thickness must be greater than 400 µ
* absence of corneal scarring
* patients must meet the diagnostic criteria for keratoconus, which include one or more of the following features:

  * high myopia
  * corneal ectasia as viewed by slit-lamp exam or measured by pachometry
  * Vogt's striae
  * topographic findings of superior flattening and inferior steepening of the cornea
  * presence of Fleischer ring

Exclusion Criteria:

* history of prior ocular surgery (history of contact lens use is not an exclusion criterion)
* average corneal power > 60 D
* presence of corneal scarring
* corneal thickness 400 µ or less
* history of herpes simplex virus keratitis
* history of uveitis
* pre-existing glaucoma

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 24 months
Spherical equivalent power of the cornea (Best spectacle refraction) | 24 months
KMax: the maximum corneal curvature | 24 months
Average corneal power of the cornea in the central 4 mm. | 24 months

SECONDARY OUTCOMES:
Corneal resistance factor. | 24 months
Maximal posterior surface elevation of the cornea. | 24 months
Apical corneal thickness. | 24 months
Endothelial count. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James J Reidy, M.D., Principal Investigator — SUNY at Buffalo School of Medicine & Biomedical Sciences
Locations (2):
- United States (2):
  - Fichte,Endl, & Elmer EyeCare, Amherst, New York
  - The Ira G. Ross Eye Institute, Buffalo, New York

REFERENCES:
- [Result] Natarajan R, Padmanabhan P, Guruswami S. Hydration behavior of porcine cornea crosslinked with riboflavin and ultraviolet A. J Cataract Refract Surg. 2007 Sep;33(9):1503. doi: 10.1016/j.jcrs.2007.04.047. No abstract available. PMID 17720054
- [Result] Mazzotta C, Balestrazzi A, Traversi C, Baiocchi S, Caporossi T, Tommasi C, Caporossi A. Treatment of progressive keratoconus by riboflavin-UVA-induced cross-linking of corneal collagen: ultrastructural analysis by Heidelberg Retinal Tomograph II in vivo confocal microscopy in humans. Cornea. 2007 May;26(4):390-7. doi: 10.1097/ICO.0b013e318030df5a. PMID 17457184
- [Result] Spoerl E, Mrochen M, Sliney D, Trokel S, Seiler T. Safety of UVA-riboflavin cross-linking of the cornea. Cornea. 2007 May;26(4):385-9. doi: 10.1097/ICO.0b013e3180334f78. PMID 17457183
- [Result] Mazzotta C, Traversi C, Baiocchi S, Sergio P, Caporossi T, Caporossi A. Conservative treatment of keratoconus by riboflavin-uva-induced cross-linking of corneal collagen: qualitative investigation. Eur J Ophthalmol. 2006 Jul-Aug;16(4):530-5. doi: 10.1177/112067210601600405. PMID 16952090
- [Result] Wollensak G. Crosslinking treatment of progressive keratoconus: new hope. Curr Opin Ophthalmol. 2006 Aug;17(4):356-60. doi: 10.1097/01.icu.0000233954.86723.25. PMID 16900027
- [Result] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- [Result] Kohlhaas M, Spoerl E, Schilde T, Unger G, Wittig C, Pillunat LE. Biomechanical evidence of the distribution of cross-links in corneas treated with riboflavin and ultraviolet A light. J Cataract Refract Surg. 2006 Feb;32(2):279-83. doi: 10.1016/j.jcrs.2005.12.092. PMID 16565005
- [Result] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Result] Mencucci R, Mazzotta C, Rossi F, Ponchietti C, Pini R, Baiocchi S, Caporossi A, Menchini U. Riboflavin and ultraviolet A collagen crosslinking: in vivo thermographic analysis of the corneal surface. J Cataract Refract Surg. 2007 Jun;33(6):1005-8. doi: 10.1016/j.jcrs.2007.03.021. PMID 17531694
- See also: National Keratoconus Foundation — http://www.nkcf.org